CLINICAL TRIAL: NCT05456282
Title: Acute Effects of Automated Mechanical Peripheral Stimulation on Cardiovascular, Functional Capacity and Postural Control in Patients With Parkinson's Disease
Brief Title: Acute Effects of AMPS on Cardiovascular, Functional Capacity and Postural Control in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Antonio Roberto Zamunér, Adjunct Professor, Universidad Católica del Maule
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 11180310
Record Dates: First submitted 2022-07-04; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants will randomly assigned to receive one of two alternative interventions (SHAM or AMPS) in the first session and the other intervention during the second visit. Participants will be assessed before and after each session.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMPS first, then SHAM (Experimental): Participants will receive first one session of automated mechanical peripheral stimulation (AMPS) with intensity at the pain threshold. Then, after a 2-week washout, they will receive one session of a simulated automated mechanical peripheral stimulation (SHAM) with intensity at the sensory threshold.
  Interventions: Device: Automated mechanical peripheral stimulation; Device: SHAM
- SHAM first, then AMPS (Sham Comparator): Participants will receive first one session of simulated automated mechanical peripheral stimulation (SHAM) with intensity at the sensory threshold. Then, after a 2-week washout, they will receive one session of automated mechanical peripheral stimulation (AMPS) with intensity at the pain threshold.
  Interventions: Device: Automated mechanical peripheral stimulation; Device: SHAM

INTERVENTIONS:
Device: Automated mechanical peripheral stimulation — Automated mechanical pressure reaching the pain threshold in four specific points at the foots soles
  Other Names: Mechanical somatosensory stimulation; Gondola
Device: SHAM — Automated mechanical pressure reaching the sensory threshold in four specific points at the foots soles

SUMMARY:
Considering that Parkinson's Disease (PD) can significantly compromise functional mobility and cardiovascular system in patients with PD, therapies aimed at improving these aspects, mainly by non-pharmacological and non-invasive methods, are paramount. This clinical trial will study the acute effects of plantar stimulation using a therapy called automated peripheral mechanical stimulation (AMPS) on cardiovascular and functional mobility in patients with PD.

The hypothesis of this study is that one single session will be effective in improving, acutely, the cardiovascular system and functional capacity in patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's disease
* Scoring 1 to 3 on the Hoehn and Yhar scale
* Pharmacological treatment unchanged for at least 30 days prior the study

Exclusion Criteria:

* Signs of cognitive decline, based on the results of the Mini Mental State Examination
* Cardiorespiratory, neuromuscular and musculoskeletal diseases not related to PD
* Sensory peripheral neuropathy, diabetes or any other disease known to promote autonomic dysfunction

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Timed up and go | 1 hour
  Time spent for the participant to rise from a standard chair without armrests, walk 3 meters straight at their preferred speed, turn, walk back to the chair and sit down again. Participants will perform the test twice and the lowest total duration will be considered as the outcome. The outcome measure is assessed as a difference or change from baseline to immediately after the intervention (about 1 hour from baseline assessment).
Center of Pressure | 1 hour
  Stabilometric variables of the center of pressure assessed using a 3D Force Plate (Kistler, US). Outcomes include anteroposterior and mediolateral velocity, root mean square and area) of the center of pressure. The outcome measure is assessed as a difference or change from baseline to immediately after the intervention (about 1 hour from baseline assessment).
Heart rate variability | 1 hour
  R-R intervals (time between every electrocardiogram R waves) will be recorded using a Polar V800 (Polar Electro Oy, Finland) and its variability will be quantified using linear and nonlinear methods. The outcome measure is assessed as a difference or change from baseline to immediately after the intervention (about 1 hour from baseline assessment).

SECONDARY OUTCOMES:
Tinetti Test | 1 hour
  Participants will be asked to: 1) firmly sit on a chair without armrests for at least 10 s; 2) stand up freely and keep the position for at least 10 s; 3) close the eyes during orthostatic position for at least 5 s; 4) control balance keeping the eyes closed while nudged by the clinician; 5) open the eyes and maintain upright position for at least 10 s; 6) perform a 360º turn around himself/herself; 7) sit down on the chair; and 8) walk as straight as possible for at least 10 m. The Tinetti test total score ranges from 0 to 28. The lower the score on the Tinetti test, the lower the functional mobility and the higher the risk of falling. The outcome measure is assessed as a difference or change from baseline to immediately after the intervention (about 1 hour from baseline assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio R Zamunér, PhD, Principal Investigator — Universidad Católica del Maule
Locations (1):
- Universidad Católica del Maule - Campus San Miguel, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: No
Participant data will be shared upon request at the end of the study.